CLINICAL TRIAL: NCT06764459
Title: Molecular Characterization of Patients With Acute Myeloid Leukemia and the Impact of Clonal Evolution in the Response to Therapeutic Treatments
Acronym: CLEV-LAM-2022
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CLEV-LAM-2022; RC-2022-2773282 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Myeloid Leukemia, Acute
Keywords: AML; FLT3; single cell sequencing
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to analyze patients with mutated FLT3 AML treated with specific therapy by means of molecular characterization methods, to identify the presence of clones and subclones at onset and to be able to follow their evolution during therapeutic treatment.

DETAILED DESCRIPTION:
This study aims to analyze patients with mutated FLT3 AML treated with specific therapy by means of single-cell molecular characterization methods, to identify the presence of clones and subclones at onset and to be able to follow their evolution during therapeutic treatment. In this way, it is possible to study how the mutational profile varies under therapeutic pressure and identify any alterations responsible for resistance. It will thus be possible to define a panel of new molecular markers to be included in the diagnostic routine to identify early patients refractory/resistant to treatment with FLT3 inhibitors and thus improve the therapeutic approach of these patients.

ELIGIBILITY:
Inclusion Criteria:

* FLT3 mutated

Exclusion Criteria:

* Respoder to therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Flt3 mutated patients treated with specific inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Refractoriness to therapy | At the end of the enrollment 3 years
  Selected patients, as they are mutated in FLT3, following therapy with specific inhibitors must show refractoriness to treatment in order to continue the study and investigate in single cell the presence of clones or subclones responsible for any relapses.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Ottaviani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico di Sant'Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided